CLINICAL TRIAL: NCT03536494
Title: Effectiveness of a Structured Intervention to Optimize Both the Use of Mirabegron, a β3 Receptor Agonist, and Facilitate Its Discontinuation: a Quasi-experimental Study
Brief Title: Effectiveness of a Structured Intervention to Optimize the Use of Mirabegron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catalan Institute of Health (Other Government)
Responsible Party: Principal Investigator, Eladio Fernandez Liz, Principal Investigator, Catalan Institute of Health
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ICS-MIR-2018-01
Record Dates: First submitted 2018-04-23; First posted 2018-05-24 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive bladder; Mirabegron; Persistence; Patient-Centered Care; Inappropriate prescribing; Discontinuation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Intervention group: Patients with mirabegron prescription from 1st January 2017 to 31st December 2017 assigned to any of the 17 urban primary health care centers located in the northern area of Barcelona belong to the Catalan Institute of Health (CIH).
  Control group (CG): All the other patients with mirabegron prescription assigned to any of the other 34 PHC located in Barcelona belonging to the CIH.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirabegron intervention (Experimental): Review the use of mirabegron and its discontinuation
  Interventions: Behavioral: Review the use of mirabegron and its discontinuation
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Review the use of mirabegron and its discontinuation — A structured intervention was designed consisting of four major sections:
  * General practitioners: information and training with written material and patient-centred prescribing.
  * Specialized hospital care: information regarding the intervention for urologists and gynaecologists.
  * Management support with the definition of a structured strategy.
  * Monthly monitoring of the intervention.
  Arms: Mirabegron intervention

SUMMARY:
This study was a multicentre, quasi-experimental design, controlled, before-and-after trial to estimate the effectiveness related to the review of mirabegron use and, if appropriate, its discontinuation.

Intervention group: Patients with mirabegron prescription assigned to any of the 17 primary health care centers (PHC) located in the northern area of Barcelona.

Control group: All the other patients assigned to any of the other 34 health care centers in Barcelona belonging to the Catalan Institut of Health (CIH).

The structured intervention included initiatives with general practitioners and urologists/gynaecologists, management support from health care authorities, and monthly feed-back monitoring to general practitioners (GPs).

The follow-up period was 12 months, from January 1st to December 31st, 2017.

DETAILED DESCRIPTION:
A quasi-experimental design with before/after measurement and a control group was used.

The objective was to identify the effectiveness of a training activity on the review of treatments. In addition, it was proposed to establish the duration of medication in real clinical practice, and its prevalence of use before and after the intervention.

Control group: Usual care

Intervention:

* Initiatives for healthcare professionals: information and training with written material, in an diagram format, distributed to all general practitioners.
* Initiatives for specialized hospital care: information regarding the intervention for urologists and gynaecologists.
* Management support with the definition of a structured strategy for all the addresses of the PHC and GPs.
* Monthly monitoring of the intervention (feed-back to all GPs).

The intervention consisted of: a) meetings with all the directors of the PHC; b) informative meetings and sessions in the PHC; c) distribution of the diagram to all the GPs; d) lists of patients with treatment provided periodically from the medication area; and e) review of the treatments by the GPs.

If considered appropriate, and with the consent of the patient, the medication was withdrawn.

A pharmacist and a clinical pharmacologist acted as consultants in case of any doubts regarding specific patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with mirabegron prescription. The prescription could be performed by a hospital or primary care doctor.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1932 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the number of participants with treatment | Data will be collected prospectively at five points in time: Day 0; Month 3 after inclusion; Month 6 after inclusion; Month 9 after inclusion; Month 12 after inclusion
  The percentage of change from baseline of the number of participants with treatment at 3, 6, 9 and 12 months with respect to basal values (day 0)

SECONDARY OUTCOMES:
Change from baseline of the duration of treatment at 3, 6, 9, and 12 months with respect to basal values (day 0) | Data will be collected prospectively at five points in time: Day 0; Month 3 after inclusion; Month 6 after inclusion; Month 9 after inclusion; Month 12 after inclusion
  Time from treatment commencement to discontinuation in real clinical practice
Prevalence of patients with treatment | Data will be collected prospectively at two points in time: Day 0, Month 12 after inclusion
  Number of participants with treatment before and after the intervention per 1000 patients >64 years of age attended in 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eladio Fernández-Liz, PhD, Principal Investigator — Pharmacist; Pedro Vivó Tristante, Physician, Study Director — Director. Primary Health Care Center Montcada i Reixac; Antonio Aranzana Martínez, Physician, Study Chair — Director. Primary Health Care Center Rio de Janeiro; Mª Estrella Barceló Colomer, Physician, Study Chair — Clinical Pharmacologist; José Ossó Rebull, Physician, Study Chair — Director. Primary Health Care Center Sant Andreu; María José López-Dolcet, Physician, Study Chair — Director. Primary Health Care Center Service Muntanya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Result] Reeve E, Gnjidic D, Long J, Hilmer S. A systematic review of the emerging de fi nition of 'deprescribing' with network analysis: implications for future research and clinical practice. Br J Clin Pharmacol. 2015 Dec;80(6):1254-68. doi: 10.1111/bcp.12732. PMID 27006985
- [Result] Scott IA, Hilmer SN, Reeve E, Potter K, Le Couteur D, Rigby D, Gnjidic D, Del Mar CB, Roughead EE, Page A, Jansen J, Martin JH. Reducing inappropriate polypharmacy: the process of deprescribing. JAMA Intern Med. 2015 May;175(5):827-34. doi: 10.1001/jamainternmed.2015.0324. PMID 25798731
- [Result] Wagg A, Franks B, Ramos B, Berner T. Persistence and adherence with the new beta-3 receptor agonist, mirabegron, versus antimuscarinics in overactive bladder: Early experience in Canada. Can Urol Assoc J. 2015 Sep-Oct;9(9-10):343-50. doi: 10.5489/cuaj.3098. PMID 26644809
- [Result] Chapple CR, Cruz F, Deffieux X, Milani AL, Arlandis S, Artibani W, Bauer RM, Burkhard F, Cardozo L, Castro-Diaz D, Cornu JN, Deprest J, Gunnemann A, Gyhagen M, Heesakkers J, Koelbl H, MacNeil S, Naumann G, Roovers JWR, Salvatore S, Sievert KD, Tarcan T, Van der Aa F, Montorsi F, Wirth M, Abdel-Fattah M. Consensus Statement of the European Urology Association and the European Urogynaecological Association on the Use of Implanted Materials for Treating Pelvic Organ Prolapse and Stress Urinary Incontinence. Eur Urol. 2017 Sep;72(3):424-431. doi: 10.1016/j.eururo.2017.03.048. Epub 2017 Apr 14. PMID 28413126
- [Result] Wagg AS, Foley S, Peters J, Nazir J, Kool-Houweling L, Scrine L. Persistence and adherence with mirabegron vs antimuscarinics in overactive bladder: Retrospective analysis of a UK General Practice prescription database. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.12996. Epub 2017 Sep 14. PMID 28906080
- [Result] Duckett J, Balachandran A. Tolerability and persistence in a large, prospective case series of women prescribed mirabegron. Int Urogynecol J. 2016 Aug;27(8):1163-7. doi: 10.1007/s00192-016-2945-4. Epub 2016 Jan 23. PMID 26803838